CLINICAL TRIAL: NCT00705250
Title: A Phase II Study of Bendamustine HCL in Relapsed and Primary Refractory Hodgkin Lymphoma.
Brief Title: Bendamustine HCL in Relapsed and Primary Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cephalon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-041
Record Dates: First submitted 2008-06-24; First posted 2008-06-26 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Hodgkin's Disease; Lymphoma
Keywords: Bendamustine HCL
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Bendamustine Hydrochloride

ARMS (1):
- 1 (Experimental): bendamustine hcl 120mg/m^2
  Interventions: Drug: bendamustine hcl

INTERVENTIONS:
Drug: bendamustine hcl — Patients will receive bendamustine 120mg/m^2, administered as a 30-minute infusion, for two consecutive days. Cycles will be repeated every four weeks and a total of 6 cycles will be planned. Patients will receive pegfilgrastim with each cycle. Treatment will be delayed until the absolute neutrophil count is > 1000/ul and the platelet count is > 75,000/ul.

SUMMARY:
The standard treatment for patients with HL that has not responded to treatment or has come back after treatment is stem cell transplant. When patients are not eligible for transplant or when HL comes back after transplant, there are no standard treatment options. These patients can receive chemotherapy or participate in clinical trials. Bendamustine HCl is a chemotherapy agent that is effective in treating patients with various diseases, including non-Hodgkin's lymphoma, multiple myeloma, and breast cancer. It was recently approved for the treatment of chronic lymphocytic leukemia. In addition, small studies from Eastern Europe have shown that bendamustine HCl is likely effective for treating HL. This study will find out the effect of bendamustine HCl for transplant-ineligible patients with HL that has not responded to or has come back after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of Classical Hodgkin lymphoma, confirmed by the department of hematopathology at MSKCC. Patients who have relapsed after an autologous stem cell transplant must have a biopsy after transplant to confirm relapsed Hodgkin's disease. Patients who have relapsed after an allogeneic transplant must also have a biopsy posttransplant.
* Age > or = to 18
* All patients must have PET avid measurable disease.
* Last chemotherapy > or = to 4 weeks from the start of Bendamustine HCl
* Receiving no other treatment for HL
* Patients must have normal baseline cardiac function based upon echocardiogram or gated blood pool scan (MUGA) with an ejection fraction > or = to 50%
* Patients must have a serum creatinine of < or = to 1.5 mg/dl; if creatinine >1.5 mg/dl creatinine clearance must be >60 ml/minute.
* Patients must have ANC>1000/mcl and Platelets>100,000/mcl.
* Patients must have a bilirubin level of < 2.0 mg/dl in the absence of a history of Gilbert's disease (or pattern consistent with Gilbert's).
* Patients must be Hepatitis B surface antigen and Hepatitis B core antibody negative and Hepatitis C negative.
* Patients must have failed an autologous stem cell transplant or be ineligible for an autologous stem cell transplant due to chemo-refractory disease(as defined as <50% response to standard salvage chemotherapy).
* Women who are pre-menopausal must have a negative pregnancy test
* Subjects must agree to use appropriate contraception until 4 weeks after the completion of chemotherapy.
* Patients must be HIV negative.
* If patients have a history of malignancy other than cutaneous basal cell or squamous cell carcinoma, they must be disease-free for ≥ 5 years at the time of enrollment.
* Patients or their guardians must be capable of providing informed consent.

Exclusion Criteria:

* Patients with either parenchymal brain or lepto-meningeal involvement.
* 7 or more consecutive days of prednisone therapy prior to therapy.
* Known pregnancy or breast-feeding.
* Medical illness unrelated to HL, which in the opinion of the attending physician and principal investigator will preclude administration of chemotherapy safely. This includes patients with uncontrolled infection, chronic renal insufficiency, myocardial infarction within the past 6 months, unstable angina, cardiac arrhythmias other than chronic atrial fibrillation and chronic active or persistent hepatitis
* History of any malignancy for which the disease-free interval is <5 years, excluding curatively treated cutaneous basal cell or squamous cell carcinoma and carcinoma in-situ of the cervix.
* Relapse <6 months post allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Moskowitz AJ, Hamlin PA Jr, Perales MA, Gerecitano J, Horwitz SM, Matasar MJ, Noy A, Palomba ML, Portlock CS, Straus DJ, Graustein T, Zelenetz AD, Moskowitz CH. Phase II study of bendamustine in relapsed and refractory Hodgkin lymphoma. J Clin Oncol. 2013 Feb 1;31(4):456-60. doi: 10.1200/JCO.2012.45.3308. Epub 2012 Dec 17. PMID 23248254
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Patients will receive bendamustine 120mg/m2, administered as a 30-minute infusion.
Period: Overall Study
Arm/Group | All Participants
Started | 36
Completed | 34
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Patient died in car accident | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 36
Age, Continuous [Median (Full Range); unit: years] | 34 [21 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Determine the Overall Response Rate (RR) to Bendamustine HCL in Patients With Relapsed and Primary Refractory HL.
Description: The percentage of evaluable participants who achieved either a complete response (CR) or partial response (PR). CR Disappearance of all evidence of disease. (a) FDGavid or PET positive prior to therapy; mass of any size permitted if PET negative (b) Variably FDG-avid or PET negative; regression to normal size on CT. PR Regression of measurable disease and no new sites. > or = to 50% decrease in SPD of up to 6 largest dominant masses; no increase in size of other nodes (a) FDG-avid or PET positive prior to therapy; one or more PET positive at previously involved site (b) Variably FDG-avid or PET negative; regression on CT.
Time Frame: up to 3 years
Measure: Number; unit: percentage of evaluable participants
Arm/Group | All Participants
Number analyzed (Participants) | 34
percentage of evaluable participants | 56

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 5/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=36)
Febrile neutropenia (General disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Self-limited Gross Hematuria (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=36)
Thrombocytopenia (Blood and lymphatic system disorders) | 18
Anemia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 3
Fatigue (General disorders) | 30
Nausea (Gastrointestinal disorders) | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Fever (General disorders) | 4
Pneumonia (General disorders) | 4
Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Mucositis (Gastrointestinal disorders) | 2
Febrile Neutropenia (General disorders) | 2
Hematuria (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes